CLINICAL TRIAL: NCT03539666
Title: The Effect of Pork and Chicken Diets on Gut Microbiota Composition and Metabolites Related to Cardiometabolic Wellbeing
Brief Title: Effect of Diets on the Gut Microbiota Composition and Cardiometabolic Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Principal Investigator, Moul Dey, Professor, South Dakota State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRB-1804010-EXP
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Healthy
MeSH Terms: interventions — Diet; Poultry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pork (Experimental): Standard American Diet with meat source: lean pork. Diet adheres to 2015-2020 Guidelines for Americans.
  Interventions: Other: diet
- Poultry (Experimental): Standard American Diet with meat source: chicken. Diet adheres to 2015-2020 Guidelines for Americans.
  Interventions: Other: diet

INTERVENTIONS:
Other: diet — dietary patterns
  Other Names: poultry

SUMMARY:
The project will characterize human gut microbiome response to two different diets and the possible physiological and biochemical implications of such response on cardiometabolic risk factors. The study will use controlled-feeding, systems-biology, metagenomic, and metabolomic approaches to examine American dietary patterns.

DETAILED DESCRIPTION:
The study will use controlled-feeding, systems-biology, metagenomic, and metabolomic approaches to examine American dietary patterns.

ELIGIBILITY:
Inclusion Criteria:

* generally good health status based on one routine physical in the past 15 months, current health status
* normal HbA1C, weigh 110 lb or more
* Age 50 years or more, generally healthy, all races and both sexes
* generally practicing a meat-based dietary pattern, do not have any special dietary requirement, and
* willingness to comply with the study protocol, including on-site meal consumption and sample/data collection.

Exclusion Criteria:

* medication usage, probiotic, long-term antibiotic, and tobacco/drug/alcohol use
* Not on any special diet within 3 months of recruitment, and do not have any intention to lose weight.
* impaired kidney functions
* Active history of cancer, diabetes, heart, liver, and kidney diseases
* major gastrointestinal disorders in the past 3 months
* history of heart attacks or stroke
* Unable to meet in-person visit requirements for dining, picking up meals, and tests
* Any mental health condition that would affect the ability to provide written informed consent.
* If they had not had a routine health checkup during the 12 months prior to recruitment.
* If they were unwilling to abstain from taking nutritional supplements, alcohol, non-study foods, and beverage during the study period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Microbiota-dependent TMAO-response, measured as serum concentration | 10 days per diet arm
  targeted sequencing
Serum concentration of biogenic amine metabolites | 10 days per diet arm
  Metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Moul Dey, Ph.D, Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Wagner Hall 416, Brookings, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No